CLINICAL TRIAL: NCT05498584
Title: Targeting LOXL2 and Cardiac Fibrosis for Post-acute Heart Failure Treatment- A Prospective Study
Status: Recruiting | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202002486B0A3
Record Dates: First submitted 2022-08-10; First posted 2022-08-12 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2023-12

CONDITIONS: Heart Failure; With Decompensation
Keywords: heart failure; cardiac fibrosis; cardiac rehabilitation; endothelial function; cardiopulmonary exercise test; cardiac MRI
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples with less than 10 ml volume were collected from patients who had fasted overnight. The samples were then centrifuged and stored at -70°C until they were assayed to determine serum LOXL2 levels and other biomarkers. ELISA kits provided by the manufacturer (R&D Systems, Abingdon, UK) were used for analysis, following their instructions. The absorbance at 450 nm was measured using a microplate reader, and standard curves were utilized to determine cytokine levels.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Post-acute systolic heart failure patients: Patients who received at least one exercise training section within 3 months of acute heart failure discharge are placed in the CR group. Patients will receive a multi-disciplinary disease management program by a qualified HF nursing specialist. A board-certified physiatrist prescribes moderate continuous training according to a cardiopulmonary exercise test.
  Interventions: Behavioral: exercise based cardiac rehabilitation

INTERVENTIONS:
Behavioral: exercise based cardiac rehabilitation — The types of exercise are treadmill walking/walking-jogging/jogging, ergometer cycling, stair climbing, or elliptical machine training. The training intensity is gradually increased fortnightly to reach the targeted Borg's rate of perceived exertion (RPE) of 12-14. The training duration is 40 minutes, which included 5-10 minutes of warm-up and cool-down exercises. The training frequency is three sessions per week, with 36 sessions concluding a complete course.

SUMMARY:
A previous study demonstrated that a multidisciplinary cardiac rehabilitation (CR) program was associated with reduced medium- to long-term all-cause mortality in a retrospective propensity score-matched study. The investigators will further investigate the predictors including LOXl2, cardiac MRI, and endothelial function that will benefit from a successful CR.

DETAILED DESCRIPTION:
Acute heart failure (HF) is a major cause of morbidity and mortality worldwide. The Taiwan national health insurance launched HF post-acute care program with a multi-discipline treatment strategy to improve care quality and reduce the readmission rate on July 1, 2017. A previous study showed heart failure disease management program (HFDMP) is beneficial for reducing recurrent events of HF readmission, especially in the ischemic cardiomyopathy population. The key element of HFDMP is cardiac rehabilitation and exercise training. Lysyl oxidase-like 2 (LOXl2) is an enzyme, which crosslinks collagen in fibrotic processes such as liver cirrhosis, lung fibrosis, cardiac fibrosis, and heart failure. An animal study showed the correlation between cardiac fibrosis and LOXl2 serum level. In a previous clinical prospective cohort study (CMRPG8H1271), the investigators recruited 40 patients who were discharged from acute decompensated heart failure. During the follow-up period, 10 patients suffered from cardiovascular mortality. The investigators found that the LOXl2 level is higher in patients with mortality than without.

Cardiac fibrosis is characterized by systolic or diastolic dysfunction that results from the accumulation of extracellular connective tissue proteins in the heart's interstitium. Both clinical evidence and experimental studies have suggested that fibrotic changes in the heart are reversible.

The investigators hypothesize that multi-disciplinary cardiac rehabilitation could reverse cardiac fibrosis by decreasing LOXl2 levels and improving endothelial function via reversing endothelial to mesenchymal transition (EndMT). The investigators will enroll 126 post-acute HF patients in 3 years. The investigators will follow up on endothelial function, and LOXl2 level 6 months later. The investigators will also arrange cardiac MRI sequences, such as balanced steady-state free precession (SSFP) and late gadolinium enhancement (LGE) for the diagnosis of cardiac fibrosis. A cardiopulmonary exercise test will be arranged after discharge for phase II cardiac rehabilitation. The investigators will use all-cause mortality and HF hospitalization as our primary endpoint, life quality scores (KCCQ12), and peak VO2/kg as our secondary endpoint.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must give written informed consent before any assessment is performed.
2. Inpatients >= 20 years of age, male or female.
3. Patients with a diagnosis of heart failure New York Heart Association (NYHA) class II-IV with BNP >=100 pg/mL or NT-porBNP >= 400 pg/mL ( >= 900 pg/mL if concomitant atrial fibrillation)
4. Left ventricular ejection fraction <= 40% by echocardiography or other methods

Exclusion Criteria:

1. Estimated survival time < 6 months
2. Long-term bedridden for more than 3 months
3. Cannot tolerate exercise test due to muscular skeletal disorder.
4. Cannot cooperate all functional studies
5. Ventilator dependent
6. Terminal heart status
7. Family rejects to participate in this project
8. Primary severe valvular heart disease

Ages: 20 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This study has a target enrollment of 126 HF patients admitted for worsening heart failure (HF) in 3 years, based on at least one symptom of HF and at least two signs of HF, and a change in medical treatment specifically targeting acute decompensated HF. We enroll those patients with reduced ejection fraction (LVEF <=40%). Patients must be at least 20 years of age or greater, able to walk at the time of enrollment, and expected to be discharged to home.
Sampling Method: Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2022-08-25 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
all-cause mortality | up to 36 months
  Number of Participants That Had First Occurrence of the All-cause mortality

SECONDARY OUTCOMES:
HF readmission | up to 12 months
  Number of participants that had first occurrence of the HF readmission.
enothelial function improvement | up to 6 months
  changes of FMD from baseline to 6 months
Change From Baseline to Month 6 and Month 12 for the Kansas City Cardiomyopathy Questionnaire 12 (KCCQ 12) Clinical Summary Score | Baseline, Month 6 , Month 12]
  Change from baseline to Month 6 and month 12 for the Kansas City Cardiomyopathy Questionnaire short form (KCCQ12) clinical summary score. KCCQ12 is a 12-item, self-administered instrument that quantifies physical function, symptoms (frequency, severity and recent change), social function, self-efficacy and knowledge, and quality of life. KCCQ12 clinical summary score is a composite assessment of physical limitations and total symptom scores. Scores are transformed to a range of 0-100, in which higher scores reflect better health status.

CONTACTS AND LOCATIONS:
Overall Officials: Shyh-Ming Che, MD, Principal Investigator — Chang Gung Medical Foundation
Locations (1):
- Chang Gung Memorial Hospital Heart Failure Center, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided
We will discuss with other investigators about individual participant data (IPD) sharing.